CLINICAL TRIAL: NCT04775420
Title: Mean Platelet Volume (MPV) and Neutrophil to Lymphocyte Ratio (NLR) as Predictors of Spontaneous Bacterial Peritonitis in Cirrhotic Patients
Brief Title: MPV and NLR as Predictors of SBP Diagnosis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abudeif Abdelaal, MD, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-21-02-22
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Spontaneous Bacterial Peritonitis
Keywords: Spontaneous bacterial peritonitis; Mean platelet volume; Neutrophil to lymphocyte ratio
MeSH Terms: interventions — Mean Platelet Volume

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Ascetic patients without spontaneous bacterial peritonitis
  Interventions: Diagnostic Test: Measurement of mean platelet volume (MPV) and blood neutrophil to lymphocyte ratio (NLR)
- Group 2: Ascetic patients with spontaneous bacterial peritonitis
  Interventions: Diagnostic Test: Measurement of mean platelet volume (MPV) and blood neutrophil to lymphocyte ratio (NLR)

INTERVENTIONS:
Diagnostic Test: Measurement of mean platelet volume (MPV) and blood neutrophil to lymphocyte ratio (NLR) — MPV and NLR are easily accessible and inexpensive tests

SUMMARY:
The aim of the study is to investigate the clinical utility of mean platelet volume (MPV) and neutrophil to lymphocyte ratio (NLR) as diagnostic markers for spontaneous bacterial peritonitis (SBP).

ELIGIBILITY:
Inclusion Criteria:

* Decompensated liver cirrhosis ascetic patients.

Exclusion Criteria:

* Immunocompromised patients.
* Patients who had received antibiotics before hospital admission.
* Patients on anticoagulant medications, NSAIDs, or oral contraceptive drugs.
* Patients with heart failure, diabetes mellitus, hypertension, hyperlipidemia, peripheral vascular disease, hematological disorders, and neoplastic disorders and patients with clinically overt hypothyroidism or hyperthyroidism or with clinically and laboratory-evident autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ascites due to decompensated liver cirrhosis admitted at the inpatient section of Tropical Medicine and Gastroenterology Department, Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The utility of MPV as non-invasive predictor of SBP | 1 year
  It will be measured from CBC
The utility of NLR as non-invasive predictor of SBP | 1 year
  It will be measured from CBC

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No